CLINICAL TRIAL: NCT06638229
Title: Investigation of the Effectiveness of Electrotherapy Treatment for the Spine in Individuals with Chronic Low Back Pain
Brief Title: Effectiveness of Electrotherapy Treatment in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ulger, Head of Spine Health Unit, Principal Investigator, Clinical Professor, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUSpine017
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; electrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- StimaWell (Experimental): Participants in the StimaWELL group had previously received electrotherapy treatment for the entire spine for 4 weeks, 2 days a week. Before the treatment, participants were informed about their medical condition and the planned treatment. The StimaWELL 120MTRS system (StimaWELL® 120MTRS; Schwa-medico, Wetzlarer Straße 41-43, 35630 Ehringshausen, Germany) was used for the treatment and a stimulation mat was used to apply electrical stimulation along the entire back. The 12 channels of the mat provided different current intensities to different areas and the system offered programs tailored to various therapeutic goals.
  Interventions: Device: The StimaWELL 120MTRS system
- Waitlist (No Intervention): Patients presenting to the clinic for treatment and waiting without intervention in the waitlist group after routine evaluation.

INTERVENTIONS:
Device: The StimaWELL 120MTRS system — A standardized current (dynamic deep wave stimulation) was applied to all patients. Additionally, the mat, which reached a temperature of 40°C, provided heat therapy with electrical stimulation
  Arms: StimaWell

SUMMARY:
This study investigates the effectiveness of a specific electrotherapy treatment for individuals with chronic non-specific low back pain. The participants, who had low back pain for more than three months, were divided into two groups: a treatment group and a waitlist control group. The treatment group received electrotherapy using the StimaWELL 120MTRS system, which provided electrical stimulation and heat therapy to the entire spine over four weeks. The study assessed various outcomes, including pain levels, disability, and quality of life, before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,
* LBP for more than three months,
* Pain of 3 or more according to the Numeric Pain Scale
* being literate

Exclusion Criteria:

* having a pacemaker,
* body mass index greater than 30,
* pathologies of the cervical or lumbar region,
* cervical radiculopathy, thoracic outlet syndrome, malignant conditions,
* systemic diseases, such as neurological, psychological, cardiovascular or rheumatologic conditions, loss of function due to these diseases,
* history of surgery on the spine or upper extremities,
* acute infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale | Before and after 4 weeks of treatment
  Participants' pain catastrophizing levels were measured using the Pain Catastrophizing Scale (PCS). The total score of the PCS is 52, with higher scores indicating higher levels of catastrophizing behavior.

SECONDARY OUTCOMES:
Numeric Pain Scale | Before and after 4 weeks of treatment
  Pain intensity during activity, at rest and at night was assessed with the Numeric Pain Scale. It was graded with "0" representing "no pain" and "10" representing "the worst pain imaginable".
Oswestry Disability Index | Before and after 4 weeks of treatment
  Disability level was assessed with the Oswestry Disability Index. The scale consists of 10 items, each ranging from 0 to 5, with a total score of 100. Higher scores indicate higher levels of disability.
Nottingham Health Profile | Before and after 4 weeks of treatment
  The Nottingham Health Profile was used to assess participants' health-related quality of life. The first part of the NHP contains 38 items covering six domains: pain, physical activity, emotional reactions, energy, social isolation and sleep. Each domain is scored from 0 to 100 and the total score is the sum of these domain scores. Only the first part of the NHP was used for this study

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ülger, professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided